CLINICAL TRIAL: NCT05086198
Title: Differential Effectiveness of Two Recovery Strategies at Work, Based on Mindfulness and Physical Exercise, on Levels of Job Stress A Randomized Controlled Trial
Brief Title: Two Recovery Strategies at Work, Based on Mindfulness and Physical Exercise, on Levels of Job Stress
Acronym: ERME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: Universidad Rey Juan Carlos (Other); Universidad de Zaragoza (Other); Ministerio de Ciencia e Innovación, Spain (Other Government)
Responsible Party: Principal Investigator, Miguel Ángel Santed Germán, PhD, Clinical Psychologist and Professor, Universidad Nacional de Educación a Distancia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PID2019-110490RB-I00 (1)
Record Dates: First submitted 2021-09-28; First posted 2021-10-20 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Wellness
Keywords: mindfulness; physical exercise; meditation; mental health; stress; recovery; positive and negative affect; work performance; affective job satisfaction
MeSH Terms: conditions — Motor Activity; Psychological Well-Being | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial of three groups is proposed, with pretest, posttest and four follow-ups at 1, 2, 3 and 6 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of trial participants and care providers is not possible because of obvious differences between the interventions. However, participants will be blinded in terms of which intervention is considered the experimental one.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-based intervention (MBI) (Experimental): A 8-week mindfulness-based intervention. From 15 to 30 minutes of practice per session, three times/week through audio guided meditations.
  Interventions: Behavioral: Mindfulness-based intervention
- Physical exercise (PE) (Active Comparator): A 8-week physical exercise intervention. From 15 to 30 minutes of practice per session, three times/week through workout videos.
  Interventions: Behavioral: Physical exercise
- Wait list (WL) (No Intervention): The participants will continue their work activity as usual. This arm will receive one of the two previous interventions once the study finished.

INTERVENTIONS:
Behavioral: Mindfulness-based intervention — An instructor trained in Mindfulness-based Stress Reduction (MBSR; Kabat-Zinn, 1990) will conduct meditations lasting 15 to 30 minutes. The participants will have a mobile application designed ad hoc with the practice of the week so they can do it individually at home.
  Arms: Mindfulness-based intervention (MBI)
Behavioral: Physical exercise — An aerobic and fitness trainer will conduct aerobic exercise lasting 15 to 30 minutes. The participants will watch it in a video platform. They will not be able to do anaerobic exercise like weight lifting. The intensity of the chosen exercise will be moderate, maintaining between 120-140 beats per minute.
  Arms: Physical exercise (PE)

SUMMARY:
The present study aims to compare the differential effects of a mindfulness-based intervention (MBI) and physical exercise (PE) on different stress and health variables by self-reports. A randomized controlled trial of three groups is proposed, with pretest, posttest and four follow-ups at 1, 2, 3 and 6 months that would be developed among the employees of two large multinationals.

DETAILED DESCRIPTION:
Work and workplace related problems are common sources of stress. Work-related stress is associated with a decrease in productivity, greater absenteeism, accidents and injuries, mental illness, greater errors, and poor performance, among others, which involve significant financial costs. Therefore, it is crucial to find coping strategies that are effective in reducing such stress. Probably, the most appropriate strategies, for their real possibilities of implementation, for their easy execution, low cost and for the empirical support they have, are mindfulness-based interventions (MBIs) and physical exercise (PE). Both types of practices have shown beneficial effects for physical health, mental health and psychological well-being in general. Different investigations have compared the implementation of MBI and PE, both combined and separately, with interesting results.

The main objective is to evaluate the interactive effects of group x time, the intragroup changes and the differences between groups, in the different moments (pretest, posttest, 1, 2, 3 and 6-months follow-up) on general health, stress, affective job satisfaction, recovery, work performance, and positive and negative affect in the three groups considered; an MBI, an aerobic PE program and an inactive control / waiting list (LE) condition will be contrasted.

The secondary objective is to evaluate the trend and linear patterns in the change trajectory in the three groups during the eight weeks of intervention on fatigue, psychological distancing, sleep, work stress, and attention.

A randomized controlled trial of three groups is proposed, with pretest, posttest and four follow-ups at 1, 2, 3 and 6 months that would be developed among the employees of two large multinationals (N ≥ 150).

The primary dependent variables considered are: 1) recovery experiences; 2) perceived stress; 3) general health; 4) affective job satisfaction; 5) individual work performance; and 6) positive and negative affects. The secondary dependent variables considered are daily states of: 1) fatigue, 2) psychological distancing, 3) quality of sleep; 4) work stress; and 5) attention.

Sociodemographic data will be collected at baseline (age, gender, level of education, number of economically dependent persons, type of contract, type of working day (split/continuous), workstation type, seniority in the organization, seniority in current position and teleworking modality).

The investigators identified two candidate covariates: 1) pharmacological treatment that can influence the psychological state (measured with two alternatives, use / non-use of anxiolytics, hypnotics and other psychotropic drugs); 2) Baseline state of stress and work stress (measured using a single item scale, Likert scale from 1 to 5, 1 being very low and 5 very high)

The intervention program is structured for 8 weeks, during which the two intervention groups will carry out their recovery strategy (IBM or EF), starting and increasing the practice 5 minutes every two weeks (weeks 1 and 2, 15 minutes; weeks 3 and 4, 20 minutes; weeks 5 and 6, 25; weeks 7 and 8, 30 minutes). The control group will continue as usual. Record will be taken of recovery strategies that workers perform naturally and spontaneously, and will be compared to strategies guided by interventions, as those the investigators propose.

The investigators believe that this study is a quasi-pioneering initiative because of its theme, uses a robust methodology, and will have an important scientific-technical impact. The importance of the topic addressed in terms of health and business productivity is associated with important contributions in terms of knowledge transfer to companies and society in general.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* To be a full-time worker (≥35 hours/week).

Exclusion Criteria:

* Currently practicing any type of meditation regularly.
* Currently practicing physical activity (aerobic or anaerobic) more than once a week.
* To have a physical or mental illness that prevents moderate exercise or mindfulness practice.
* Very low self-perceived work load and responsibility levels.
* Very low self-perceived stress and work stress levels.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Change in General Health with six time points data. | Baseline, Post-treatment 8 weeks from baseline, 1-month follow-up, 2-month follow-up,3-months follow-up and 6-months follow-up
  The General Health Questionnaire (GHQ-12) consists of 12 items. It is a unidimensional measure of psychological distress. It is answered on a Likert-type scale from 1 to 4 (1 = Never and 4 = Always). The score was used to generate a total score ranging from 0 to 36.
Change in stress with six time points data. | Baseline, Post-treatment 8 weeks from baseline, 1-month follow-up, 2-month follow-up,3-months follow-up and 6-months follow-up
  A single item was used: Stress refers to a person's situation when they feel tense, restless, nervous, or anxious, or are unable to sleep at night because their mind is constantly preoccupied with work-related issues. Please indicate the extent to which you currently feel this type of stress. It has five possible responses on a Likert-type scale from 1 to 5 (being 1 nothing and 5 a lot)
Change in Affective Job Satisfaction with six time points data. | Baseline, Post-treatment 8 weeks from baseline, 1-month follow-up, 2-month follow-up,3-months follow-up and 6-months follow-up
  The Brief Index of Affective Job Satisfaction (BIAJS)-Spanish version (BIAJS) consists of 7 items. It is an overall measure of affective job satisfaction. It measures satisfaction in five facets: promotion, co-workers, work itself, supervision and salary. It is answered on a Likert-type scale from 1 to 5 (1 = Strongly disagree and 5 = Strongly agree). The score was used to generate a total score ranging from 7 to 35.
Change in Need for Recovery with six time points data. | Baseline, Post-treatment 8 weeks from baseline, 1-month follow-up, 2-month follow-up,3-months follow-up and 6-months follow-up
  The Need for Recovery (NFR) Scale consists of 9 items. It facilitates the understanding of the factors that can lead to sustainable working and employability. It is answered on a Likert-type scale from 1 to 5 (1 = Never and 5 = Always). The score was used to generate a total score ranging from 1 to 100.Our research team will carry the validation of the Spanish version of NFR.
Change in Individual Work Performance with six time points data. | Baseline, Post-treatment 8 weeks from baseline, 1-month follow-up, 2-month follow-up,3-months follow-up and 6-months follow-up
  The Individual Work Performance Questionnaire (IWPQ)-Brief Spanish version (IWPQ) has 18 items. It measures the three main dimensions of job performance: task performance, contextual performance, and counterproductive work behavior. It is answered on a Likert-type scale from 1 to 5 (1 = Never or Seldom and 5 = Always or Often). The score was used to generate a total score ranging from 18 to 90.
Change in Positive and Negative Affect with six time points data. | Baseline, Post-treatment 8 weeks from baseline, 1-month follow-up, 2-month follow-up,3-months follow-up and 6-months follow-up
  The PANAS Scales of Positive and Negative Affect (PANAS) - Spanish version has 20 items. It is the most widely used scale of affectivity. It has two dominant dimensions, positive affect (10 items) and negative affect (10 items) It is answered on a Likert-type scale from 1 to 5 (1 = Very slightly or Not at all and 5 = Extremely). The score was used to generate a total score ranging from 20 to 100.

SECONDARY OUTCOMES:
Change in Fatigue (single-item measure from the Single-Item Fatigue Measure). | 4 days per week during the 8-week interventions
  Single-Item on fatigue level:" Indicate what level of fatigue you felt today". The response is rcorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Psychological distancing (item n. 3 from the Recovery Experience Questionnaire). | 4 days per week during the 8-week interventions
  Single-Item on Psychological distancing level: "After work, I have been able to "disconnect". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Sleep (item n. 6 from the Pittsburg Sleep Quality Index). | 4 days per week during the 8-week interventions
  Single-Item on Sleep: "How did you sleep last night?". The responses are articulated on a Likert-type scale from 1 to 5 (1 = very bad and 5 = very good)
Change in Work stress (single-item measure from the Single-item Measure of Stress Symptoms). | 4 days per week during the 8-week interventions
  Single-Item on work stress: "Indicate the extent to which you have felt stressed, tense, nervous, or anxious today". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".
Change in Mindfulness (item n. 3 from the Five Facets Mindfulness Questionnaire). | 4 days per week during the 8-week interventions
  Single-Item on attention: "Today it has been difficult for me to be attentive to what required my attention at all times". The response is recorded on a 5-point Likert scale varying from "not at all" to "very much".

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Santed, PhD, Principal Investigator — UNED
Locations (1):
- Sara Cuerva Navas, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The investigators will deposit data sets associated with the research in an Institutional Research Data Repository. If that is not possible, the interested parties may contact the corresponding author of the articles who will provide them with the required information.

REFERENCES:
- [Background] Sharma M, Rush SE. Mindfulness-based stress reduction as a stress management intervention for healthy individuals: a systematic review. J Evid Based Complementary Altern Med. 2014 Oct;19(4):271-86. doi: 10.1177/2156587214543143. Epub 2014 Jul 22. PMID 25053754
- [Background] Geurts SA, Sonnentag S. Recovery as an explanatory mechanism in the relation between acute stress reactions and chronic health impairment. Scand J Work Environ Health. 2006 Dec;32(6):482-92. doi: 10.5271/sjweh.1053. PMID 17173204
- [Background] Goyal M, Singh S, Sibinga EM, Gould NF, Rowland-Seymour A, Sharma R, Berger Z, Sleicher D, Maron DD, Shihab HM, Ranasinghe PD, Linn S, Saha S, Bass EB, Haythornthwaite JA. Meditation programs for psychological stress and well-being: a systematic review and meta-analysis. JAMA Intern Med. 2014 Mar;174(3):357-68. doi: 10.1001/jamainternmed.2013.13018. PMID 24395196
- [Background] Hulsheger UR, Alberts HJ, Feinholdt A, Lang JW. Benefits of mindfulness at work: the role of mindfulness in emotion regulation, emotional exhaustion, and job satisfaction. J Appl Psychol. 2013 Mar;98(2):310-25. doi: 10.1037/a0031313. Epub 2012 Dec 31. PMID 23276118
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Sonnentag S, Venz L, Casper A. Advances in recovery research: What have we learned? What should be done next? J Occup Health Psychol. 2017 Jul;22(3):365-380. doi: 10.1037/ocp0000079. Epub 2017 Mar 30. PMID 28358572
- [Background] de Bruin EI, van der Zwan JE, Bogels SM. A RCT Comparing Daily Mindfulness Meditations, Biofeedback Exercises, and Daily Physical Exercise on Attention Control, Executive Functioning, Mindful Awareness, Self-Compassion, and Worrying in Stressed Young Adults. Mindfulness (N Y). 2016;7(5):1182-1192. doi: 10.1007/s12671-016-0561-5. Epub 2016 Jul 2. PMID 27642375
- [Background] van der Zwan JE, de Vente W, Huizink AC, Bogels SM, de Bruin EI. Physical activity, mindfulness meditation, or heart rate variability biofeedback for stress reduction: a randomized controlled trial. Appl Psychophysiol Biofeedback. 2015 Dec;40(4):257-68. doi: 10.1007/s10484-015-9293-x. PMID 26111942
- [Background] Wolever RQ, Bobinet KJ, McCabe K, Mackenzie ER, Fekete E, Kusnick CA, Baime M. Effective and viable mind-body stress reduction in the workplace: a randomized controlled trial. J Occup Health Psychol. 2012 Apr;17(2):246-258. doi: 10.1037/a0027278. Epub 2012 Feb 20. PMID 22352291
- [Background] Heikkila K, Fransson EI, Nyberg ST, Zins M, Westerlund H, Westerholm P, Virtanen M, Vahtera J, Suominen S, Steptoe A, Salo P, Pentti J, Oksanen T, Nordin M, Marmot MG, Lunau T, Ladwig KH, Koskenvuo M, Knutsson A, Kittel F, Jockel KH, Goldberg M, Erbel R, Dragano N, DeBacquer D, Clays E, Casini A, Alfredsson L, Ferrie JE, Singh-Manoux A, Batty GD, Kivimaki M; IPD-Work Consortium. Job strain and health-related lifestyle: findings from an individual-participant meta-analysis of 118,000 working adults. Am J Public Health. 2013 Nov;103(11):2090-7. doi: 10.2105/AJPH.2012.301090. Epub 2013 May 16. PMID 23678931
- [Result] Carral P, Alcover CM. Measuring Age Discrimination at Work: Spanish Adaptation and Preliminary Validation of the Nordic Age Discrimination Scale (NADS). Int J Environ Res Public Health. 2019 Apr 22;16(8):1431. doi: 10.3390/ijerph16081431. PMID 31013640
- [Result] Fernandez-Munoz JJ, Topa G. Older Workers and Affective Job Satisfaction: Gender Invariance in Spain. Front Psychol. 2018 Jun 8;9:930. doi: 10.3389/fpsyg.2018.00930. eCollection 2018. PMID 29937748
- [Result] de Croon EM, Sluiter JK, Frings-Dresen MH. Psychometric properties of the Need for Recovery after work scale: test-retest reliability and sensitivity to detect change. Occup Environ Med. 2006 Mar;63(3):202-6. doi: 10.1136/oem.2004.018275. PMID 16497863
- [Result] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Elo AL, Leppanen A, Jahkola A. Validity of a single-item measure of stress symptoms. Scand J Work Environ Health. 2003 Dec;29(6):444-51. doi: 10.5271/sjweh.752. PMID 14712852
- [Result] Sonnentag S, Fritz C. The Recovery Experience Questionnaire: development and validation of a measure for assessing recuperation and unwinding from work. J Occup Health Psychol. 2007 Jul;12(3):204-21. doi: 10.1037/1076-8998.12.3.204. PMID 17638488
- [Result] van Hooff ML, Geurts SA, Kompier MA, Taris TW. "How fatigued do you currently feel?" Convergent and discriminant validity of a single-item fatigue measure. J Occup Health. 2007 May;49(3):224-34. doi: 10.1539/joh.49.224. PMID 17575403
- See also: Assessing Job Performance Using Brief Self-report Scales: The Case of the Individual Work Performance Questionnaire — https://doi.org/10.5093/jwop2019a21
- See also: PANAS scale of positive and negative affect: factor validation and cross-cultural convergence — https://dialnet.unirioja.es/servlet/articulo?codigo=2011515
- See also: Psychometric properties and normative values of the General Health Questionnaire (GHQ-12) in the general Spanish population — https://www.redalyc.org/pdf/337/33715423008.pdf
- See also: European Agency for Safety and Health at Work — https://www.europarl.europa.eu/factsheets/en/sheet/56/health-and-safety-at-work